CLINICAL TRIAL: NCT04908852
Title: A Pilot Study to Assess Feasibility and Explore Variability in Biomarkers and Patient Reported Outcome Measures in Patients Undergoing Induction Chemotherapy for Acute Myeloid Leukemia
Brief Title: Feasibility Pilot Exploring Variability in Biomarkers and PROs in AML
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Marilyn Hammer, PhD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 21-161; N98F20P00013 (Other: National Institute of Nursing Research (NINR))
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: This is a prospective, longitudinal, observational exploratory study. Ten subjects will be enrolled and will complete baseline and week 4 blood draws and symptom questionnaires at baseline, 1-, 2-, 3- and 4-weeks.
  Interventions: Other: Blood Sample Collection - Observational Study; Other: Symptom questionnaires - Observational Study

INTERVENTIONS:
Other: Blood Sample Collection - Observational Study — Blood samples will be collected at enrollment and week 4 and used in analyses to understand associations between metabolic function and symptom experiences.
Other: Symptom questionnaires - Observational Study — Symptom questionnaires at baseline, 1-, 2-, 3- and 4-weeks.

SUMMARY:
This research study is being conducted to help understand how the symptoms during treatment for acute myeloid leukemia (AML) may be affected by metabolism and how best to study this association. Symptoms include experiences like fatigue, sleep disturbance, pain, and depression.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, observational exploratory study. Ten participants will be enrolled and will complete baseline and week 4 blood sample collections. Symptom questionnaires will be completed at baseline, 1-, 2-, 3- and 4-weeks.

This research study is a Pilot Study, which means it is the first time that researchers are studying the associations between symptoms and metabolism in this way.

The National Institute of Nursing Research is supporting this research study by providing funding for the research study.

ELIGIBILITY:
Inclusion Criteria:

* The Cantor Center CRC will attend weekly protocol meetings in the DFCI adult leukemia center to identify eligible patients and will confirm eligibility by reviewing the electronic health record and, if needed, contacting the treating physician. Subjects enrolled in clinical trials or other studies requiring extra blood samples and/or completion of questionnaires will be discussed with their oncology care team and/or investigators of the other study teams to ensure avoidance of excess subject burden. Only subjects deemed appropriate for enrollment without adding excess burden will be approached about this study.
* Inclusion Criteria:

  * Adult (18+ years old)
  * New diagnosis of acute myeloid leukemia (AML)
  * Admitted to the DFCI Inpatient Hospital in the BWH for intensive induction chemotherapy (e.g., 7+3 regimen)
  * Eastern Cooperative Oncology Group Scale of Performance Status (ECOG PS) ≤ 3 OR Karnofsky Performance Status (KPS) ≥ 50
  * Ability to comprehend and speak English
  * Ability to provide informed consent

Exclusion Criteria:

* Cognitive or psychiatric conditions prohibiting study consent or participation
* Multiple primary cancers
* A treating clinician reports that the subject is inappropriate for the study or that the study presents excess subject burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with acute myeloid leukemia (AML) admitted to Dana Farber Cancer Institute for induction chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Completion rate | 30 Days
  Evaluate the feasibility of conducting this type of study on an in-patient oncology unit (i.e., >70% of enrolled participants will complete 30-day outcome assessments). Using descriptive statistics, feasibility will be calculated as the percent of eligible participants who enroll in the study and among those who enroll, the percent who complete the study. Using a 90%-exact binomial confidence interval estimate, 8 out of 10 participants completing the 30-day study will be considered acceptable for feasibility

SECONDARY OUTCOMES:
Enrollment rate | 30 Days
  Evaluate the feasibility of conducting this type of study on an in-patient oncology unit (i.e., ≥ 50% approach-to enrollment rate of eligible participants). Using descriptive statistics, feasibility will be calculated as the percent of eligible participants who enroll in the study and among those who enroll, the percent who complete the study. Using a 90%-exact binomial confidence interval estimate, 8 out of 10 participants completing the 30-day study will be considered acceptable for feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn J. Hammer, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu